CLINICAL TRIAL: NCT00045292
Title: A Phase III Multicenter Study of Cytomegalovirus Prophylaxis With Valacyclovir for the Prevention of Serious Fungal and Bacterial Infections Among Cytomegalovirus Seronegative Recipients of Cytomegalovirus Seropositive Sx Stem Cell Transplants
Brief Title: Valacyclovir in Preventing Cytomegalovirus Infection in Patients Who Are Undergoing Donor Stem Cell Transplantation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Supportive Care
Other Study IDs: 1603.00; FHCRC-1603.00; NCI-H02-0092; CDR0000256871 (Registry Identifier: PDQ)
Record Dates: First submitted 2002-09-06; First posted 2003-01-27 (Estimated); Last update posted 2010-09-21 (Estimated); Status verified 2010-09

CONDITIONS: Cancer
Keywords: infection; accelerated phase chronic myelogenous leukemia; blastic phase chronic myelogenous leukemia; childhood chronic myelogenous leukemia; chronic phase chronic myelogenous leukemia; relapsing chronic myelogenous leukemia; adult acute lymphoblastic leukemia in remission; childhood acute lymphoblastic leukemia in remission; recurrent adult acute lymphoblastic leukemia; recurrent childhood acute lymphoblastic leukemia; untreated adult acute lymphoblastic leukemia; untreated childhood acute lymphoblastic leukemia; adult acute myeloid leukemia in remission; childhood acute myeloid leukemia in remission; recurrent adult acute myeloid leukemia; recurrent childhood acute myeloid leukemia; secondary acute myeloid leukemia; untreated adult acute myeloid leukemia; untreated childhood acute myeloid leukemia and other myeloid malignancies; atypical chronic myeloid leukemia; chronic eosinophilic leukemia; chronic idiopathic myelofibrosis; chronic neutrophilic leukemia; chronic myelomonocytic leukemia; juvenile myelomonocytic leukemia; de novo myelodysplastic syndromes; myelodysplastic/myeloproliferative disease, unclassifiable; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; disseminated neuroblastoma; recurrent neuroblastoma; noncontiguous stage II adult diffuse large cell lymphoma; recurrent adult diffuse large cell lymphoma; stage III adult diffuse large cell lymphoma; stage IV adult diffuse large cell lymphoma; noncontiguous stage II adult Burkitt lymphoma; recurrent adult Burkitt lymphoma; stage III adult Burkitt lymphoma; stage IV adult Burkitt lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; recurrent adult diffuse mixed cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage IV adult diffuse mixed cell lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; recurrent adult lymphoblastic lymphoma; recurrent childhood lymphoblastic lymphoma; stage III adult lymphoblastic lymphoma; stage IV adult lymphoblastic lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; noncontiguous stage II mantle cell lymphoma; recurrent mantle cell lymphoma; stage III mantle cell lymphoma; stage IV mantle cell lymphoma; poor prognosis metastatic gestational trophoblastic tumor; previously treated childhood rhabdomyosarcoma; recurrent Wilms tumor and other childhood kidney tumors; recurrent adult Hodgkin lymphoma; recurrent/refractory childhood Hodgkin lymphoma; recurrent childhood rhabdomyosarcoma; recurrent childhood large cell lymphoma; recurrent childhood small noncleaved cell lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; recurrent mycosis fungoides/Sezary syndrome; recurrent ovarian epithelial cancer; recurrent ovarian germ cell tumor; stage II ovarian epithelial cancer; stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer; recurrent malignant testicular germ cell tumor; stage III malignant testicular germ cell tumor; refractory chronic lymphocytic leukemia; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; refractory hairy cell leukemia; refractory multiple myeloma; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer; noncontiguous stage II small lymphocytic lymphoma; noncontiguous stage II marginal zone lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage III marginal zone lymphoma; stage IV small lymphocytic lymphoma; stage IV marginal zone lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; childhood myelodysplastic syndromes
MeSH Terms: conditions — Neoplasms; Infections; Leukemia, Myeloid, Accelerated Phase; Blast Crisis; Leukemia, Myeloid, Chronic-Phase; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Pdgfra-Associated Chronic Eosinophilic Leukemia; Primary Myelofibrosis; Leukemia, Neutrophilic, Chronic; Leukemia, Myelomonocytic, Chronic; Leukemia, Myelomonocytic, Juvenile; Myeloproliferative Disorders; Neuroblastoma; Lymphoma, Large B-Cell, Diffuse; Burkitt Lymphoma; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Wilms Tumor; Hodgkin Disease; Recurrence; Dendritic Cell Sarcoma, Interdigitating; Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides; Sezary Syndrome; Carcinoma, Ovarian Epithelial; Testicular Neoplasms; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Hairy Cell; Multiple Myeloma; Breast Neoplasms; Lymphoma, B-Cell, Marginal Zone | interventions — Acyclovir; Valacyclovir

INTERVENTIONS:
Drug: acyclovir
Drug: acyclovir sodium
Drug: valacyclovir

SUMMARY:
RATIONALE: Antivirals such as valacyclovir act against viruses and may be effective in preventing cytomegalovirus. It is not yet known if valacyclovir is effective in preventing cytomegalovirus in patients undergoing stem cell transplantation.

PURPOSE: Randomized phase III trial to determine the effectiveness of valacyclovir in preventing cytomegalovirus in patients who are undergoing donor stem cell transplantation.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the occurrence of serious invasive fungal or bacterial infections during the first 270 days after transplantation in cytomegalovirus (CMV)-negative patients receiving a CMV-positive allogeneic stem cell transplantation and valacyclovir or placebo.
* Compare the occurrence of primary CMV infection within the first 100 days after transplantation in patients treated with these regimens.
* Compare the survival of these patients at 100 days and 270 days post-transplantation.
* Compare the occurrence of CMV disease at day 100 and day 270 post-transplantation in patients treated with these regimens.
* Compare the safety of these regimens in these patients.
* Correlate the presence of CMV in stem cell product with post-transplantation CMV infection in these patients.
* Determine if subclinical CMV infection results in a virus-specific immune response (humoral and cellular) in these patients.
* Compare the quality of life of patients treated with these regimens.
* Compare resource utilization (e.g., rates of hospitalization, number of days alive out of the hospital, days in the intensive care unit, days on mechanical ventilation, use of antimicrobials and filgrastim [G-CSF], and number of invasive procedures) in patients treated with these regimens.

OUTLINE: This is a randomized, double-blind, placebo-controlled, multicenter study. Patients are stratified according to participating center and type of transplantation (matched related vs mismatched/unrelated). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral valacyclovir 4 times daily beginning with transplantation conditioning (usually day -5) and continuing until day 100 after transplantation. Patients receive high-dose acyclovir, instead of valacyclovir, IV every 8 hours beginning on day -1 and continuing until oral medications are tolerated. Allogeneic stem cells are infused on day 0.
* Arm II: Patients receive oral or IV placebo on the same schedule as in arm I. Quality of life is assessed at baseline and on days 50 and 100.

Patients are followed every 2 weeks for 6 months.

PROJECTED ACCRUAL: A total of 115-230 patients (58-115 per treatment arm) will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Disease requiring one of the following types of stem cell transplantation:

  * First myeloablative allogeneic peripheral blood stem cell
  * Unrelated cord blood
  * Bone marrow

    * Related or unrelated donor
    * T-cell depleted or non-T-cell depleted
    * CD34 selected or non-selected
* Patient must be cytomegalovirus (CMV)-seronegative and donor must be CMV-seropositive
* No transplantation with nonmyeloablative regimens, including any of the following:

  * Fludarabine and total body irradiation (TBI) (2 Gy or less)
  * TBI alone (2 Gy)
  * Fludarabine, cytarabine, and idarubicin
  * Fludarabine and melphalan (140 mg/m^2 or less)
* No definite or probable pre-transplantation diagnosis of invasive mold infection (aspergillosis, fusariosis, or zygomycosis), including pulmonary or hepatic nodules consistent with invasive mold infection for which patients are receiving targeted prophylaxis with amphotericin or other mold-active products
* No pre-transplantation-CMV disease (gastrointestinal or pneumonia)

PATIENT CHARACTERISTICS:

Age

* 12 and over

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Other

* HIV negative
* No hypersensitivity to acyclovir or valacyclovir
* Not pregnant
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Disease Characteristics

Chemotherapy

* See Disease Characteristics

Endocrine therapy

* Not specified

Radiotherapy

* See Disease Characteristics

Surgery

* Not specified

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2002-04; Study Completion 2004-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Garrett Nichols, MD, MSC, Study Chair — Fred Hutchinson Cancer Center
Locations (6):
- United States (6):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Stanford Cancer Center at Stanford University Medical Center, Stanford, California
  - UNMC Eppley Cancer Center at the University of Nebraska Medical Center, Omaha, Nebraska
  - Baylor University Medical Center, Dallas, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Fred Hutchinson Cancer Research Center, Seattle, Washington